CLINICAL TRIAL: NCT05699304
Title: Complications After Thyroid Surgeries: 10 Years' Experience
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Taha Aly, Assistant Professor, South Valley University
Other Study IDs: SVU-MED-SUR011-4-22-12-515
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Thyroid
Keywords: Thyroidectomy; Hypocalcemia; Stridor; Bleeding; Recurrent Laryngeal Nerve
MeSH Terms: conditions — Thyroid Diseases; Hypocalcemia; Respiratory Sounds; Hemorrhage | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thyroidectomy — Thyroidectomy

SUMMARY:
Thyroidectomy is one of the commonest elective surgeries in surgical practice nowadays. It is associated with wide range of complications, from unnoticed events up to lifelong problems and even life-threatening complications. The most troublesome are bleeding, nerve injury and hypocalcemia. The current study was conducted to report the incidence and predictive factors for perioperative complications, aiming to point out preventive measures.

DETAILED DESCRIPTION:
All files of all patients that had thyroidectomy in the hospital in the last 10 yeas will be reviewed. All demographic and peri-operative data will be collected, tabulated and analyzed.

Incidence and pre-operative predictive factors of every single complication will pointed out and discussed.

ELIGIBILITY:
Inclusion Criteria:

* All patients had thyroid disease and performed thyroidectomy in the last 10 years in our hospital.

Exclusion Criteria:

* Uncompleted files.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients had thyroid diseases and had thyroidectomy in our hospital in last 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Recurrent Laryngeal nerve injury | 1 week
  Recurrent Laryngeal nerve injury
Bleeding | 2 days
  intraoperative or post operative bleeding.
Hypocalcemia | 6 months
  Clinically significant low serum calcium level/

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah M Taha, MD, Principal Investigator — South Valley University
Locations (1):
- Qena Faculty of Medicine, South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogbera AO, Kuku SF. Epidemiology of thyroid diseases in Africa. Indian J Endocrinol Metab. 2011 Jul;15(Suppl 2):S82-8. doi: 10.4103/2230-8210.83331. PMID 21966659
- [Background] Ernandes-Neto M, Tagliarini JV, Lopez BE, Padovani CR, Marques Mde A, Castilho EC, Mazeto GM. Factors influencing thyroidectomy complications. Braz J Otorhinolaryngol. 2012 Jun;78(3):63-9. doi: 10.1590/S1808-86942012000300012. PMID 22714849
- [Background] Zambudio AR, Rodriguez J, Riquelme J, Soria T, Canteras M, Parrilla P. Prospective study of postoperative complications after total thyroidectomy for multinodular goiters by surgeons with experience in endocrine surgery. Ann Surg. 2004 Jul;240(1):18-25. doi: 10.1097/01.sla.0000129357.58265.3c. PMID 15213613
- [Background] Khanzada TW, Samad A, Memon W, Kumar B. Post thyroidectomy complications: the Hyderabad experience. J Ayub Med Coll Abbottabad. 2010 Jan-Mar;22(1):65-8. PMID 21409907
- [Background] Potenza AS, Araujo Filho VJF, Cernea CR. Injury of the external branch of the superior laryngeal nerve in thyroid surgery. Gland Surg. 2017 Oct;6(5):552-562. doi: 10.21037/gs.2017.06.15. PMID 29142848